CLINICAL TRIAL: NCT03723590
Title: A Clinical Evaluation of an Esterified Hyaluronic Acid Matrix on Preparing Wounds in Burn Patients for Split-thickness Skin Grafting
Brief Title: A Clinical Evaluation of an Esterified Hyaluronic Acid Matrix in Burn Patients for STSG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-2018-DIV31-006
Record Dates: First submitted 2018-10-23; First posted 2018-10-29 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2021-11

CONDITIONS: Burn Wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Esterified hyaluronic acid matrix (Experimental)
  Interventions: Device: Esterified Hyaluronic Acid Matrix

INTERVENTIONS:
Device: Esterified Hyaluronic Acid Matrix — A non-woven pad composed of esterified hyaluronic acid, covered with a semipermeable silicone layer to protect the wound and control water vapor loss

SUMMARY:
Burn patients meeting inclusion criteria will receive the esterified hyaluronic acid matrix as the matrix for their wound, in conjunction with the standard of care for managing these types of wounds. The study will be divided into two phases. Phase I will entail intervention with the wound matrix and will continue until one of the following occur, sufficient granulation has occurred and the patient can receive a STSG and proceed to Phase II, the patient's physician determines an STSG is no longer necessary or two applications with the wound matrix occur and no STSG is approved. Phase II will begin following the STSG procedure. In this phase, the wound will be monitored and proportion of STSG take will be evaluated but no application of the wound matrix device will take place. This phase will continue for 28 days or if the physician deems the patient no longer needs regular care to monitor the wound, whichever occurs earlier.

ELIGIBILITY:
Inclusion Criteria:

* Has a wound originating from a thermal or electrical burn
* Target burn area is less than 20% of TBSA
* Target burn wound is greater than 0.5% of TBSA
* Patient has undergone escharectomy procedure or will undergo escharectomy on the target burn and resulting wound will likely need a split thickness skin graft, but wound site is not immediately ready for grafting
* For patients with diabetes, an A1C hemoglobin level between 11 percent (taken within 90 days)

Exclusion Criteria:

* Current active diagnosis of substance abuse, per the Investigator
* Patient currently taking non-inhaled corticosteroids
* Patient needs or is likely to need negative pressure wound therapy of the target wound after application of Hyalomatrix Wound Device
* Patient is pregnant, planning to become pregnant during study period, or breastfeeding
* Unstable medical condition as determined by the site investigator
* Patients with known sensitivities to hyaluronan, hyaluronan derivatives, silicone, or any other ingredients of the Hyalomatrix Wound Device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Esterified Hyaluronic Acid Matrix
Started | 5
Completed | 0 (Study was stopped due to business decision. Baseline information, Subject packets and data were not collected for analysis. Numbers were given based on discussion with the sites. I can change all to zero if needed.)
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Study was stopped due to business decision and baseline information, data or subject packets were not collected for analysis.
Arm/Group | Esterified Hyaluronic Acid Matrix
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Days From Initial Application of Wound Matrix to Approval of Wound to Receive a Split Thickness Skin Graft
Time Frame: Baseline to 42 days
Population: Study was stopped due to business decision and data was not collected for analysis.
Arm/Group | Esterified Hyaluronic Acid Matrix
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Wound Volume From the Time Prior to Application of the Wound Device to the Time Before the Application of STSG and After STSG
Time Frame: Baseline to 42 days
Population: Study was stopped due to business decision and data was not collected for analysis.
Arm/Group | Esterified Hyaluronic Acid Matrix
Number analyzed (Participants) | 0

3. Secondary Outcome: Length of Stay in Inpatient Unit
Time Frame: Baseline to 42 days
Population: Study was stopped due to business decision and data was not collected for analysis.
Arm/Group | Esterified Hyaluronic Acid Matrix
Number analyzed (Participants) | 0

4. Secondary Outcome: Patient Pain Rating
Time Frame: Baseline to 42 days
Population: Study was stopped due to business decision and data was not collected for analysis.
Arm/Group | Esterified Hyaluronic Acid Matrix
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Split Thickness Skin Graft Take for the Wound at 28 Days
Time Frame: 28 days
Population: Study was stopped due to business decision and data was not collected for analysis.
Arm/Group | Esterified Hyaluronic Acid Matrix
Number analyzed (Participants) | 0

6. Secondary Outcome: Proportion of Patients Who Develop an Infection of the Target Wound at Any Time Per Confirmation With Culture
Time Frame: Baseline to 70 days
Population: Study was stopped due to business decision and data was not collected for analysis.
Arm/Group | Esterified Hyaluronic Acid Matrix
Number analyzed (Participants) | 0

7. Secondary Outcome: Subject Discharge Destination
Description: The facility that the subject is discharged to will be captured.
Time Frame: Baseline to 70 days
Population: Study was stopped due to business decision and data was not collected for analysis.
Arm/Group | Esterified Hyaluronic Acid Matrix
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study stopped due to business decision. Baseline, data & Subject packets were not collected.
Description: Study stopped due to business decision. Baseline, data & Subject packets were not collected.
Arm/Group | Esterified Hyaluronic Acid Matrix
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Due to a business decision with the pandemic it was decided to terminate this study and data was never collected from the site or analyzed for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03723590/Prot_SAP_000.pdf